CLINICAL TRIAL: NCT02741375
Title: Cerebral Oximetry As an Auxiliary Diagnostic Tool in the Diagnosis of Brain Death
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Turedi, Assoc. Prof., M.D., Karadeniz Technical University
Other Study IDs: 2014/05
Record Dates: First submitted 2016-04-07; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Brain Death
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Brain Death Group (BD group): Patients assessed as brain-dead at the first clinical evaluation by the OTBD committee were definitively diagnosed with BD through repeat clinical evaluation after 24 h or through CT angiography as a corroboratory test. Patients regarded as definitely brain-dead on the basis of this evaluation were classified as the BD group.
  Interventions: Device: Somanetics 5100c (Invos oximeter cerebral/somatic Troy, MI, USA)
- Non-Brain Death Group (Non BD group): Patients assessed as brain-dead at the first clinical evaluation by the OTBD committee were definitively diagnosed with BD through repeat clinical evaluation after 24 h or through CT angiography as a corroboratory test. Patients regarded as definitely not brain-dead on the basis of this evaluation were classified as the non-BD group.
  Interventions: Device: Somanetics 5100c (Invos oximeter cerebral/somatic Troy, MI, USA)

INTERVENTIONS:
Device: Somanetics 5100c (Invos oximeter cerebral/somatic Troy, MI, USA) — All patients underwent at least 6-h NIRS monitoring using a Somanetics 5100c (Invos oximeter cerebral/somatic Troy, MI, USA) cerebral oximeter in order to determined cerebral oximetry changes.

SUMMARY:
Aim: To investigate the efficacy of cerebral oximetry (CO) as an auxiliary diagnostic tool in confirming brain death (BD).

Materials and Methods: This observational and interventional study was performed on patients with suspected BD in emergency departments and intensive care units. CO monitoring was performed for at least 6 h, and cerebral tissue oxygen saturation (ScO2) was recorded. Basal ScO2 values (basal ScO2), ScO2 values after 6 h (end ScO2), mean ScO2 values during monitoring (mean ScO2), and minimum (min ScO2) and maximum (max ScO2) ScO2 values observed during monitoring were recorded for all patients. Patients with diagnosis of BD confirmed by the organ transplantation and brain death committee were enrolled as the BD group and other patients as the non-BD group, and cerebral oxygen parameters were compared.

DETAILED DESCRIPTION:
Brain death (BD) means the irreversible loss of all brain and brain stem functions and physiopathologically the cessation of intracranial circulation. BD is a clinical diagnosis that can be made with various clinical tests. However, in order for BD to be definitely established, clinical tests performed initially need to be repeated after 24 h or to be confirmed by corroboratory tests. In addition, the obligation to confirm BD using corroboratory tests varies in current guidelines from country to country but has been eliminated except for certain specific circumstances. However, considering the adverse effects on patients awaiting donor and organ donations of the time lapse between initial and repeat tests in order to confirm BD, more rapid confirmation of definite BD is commonly made using corroboratory tests.

This study was planned with the hypothesis that this non-invasive technique using NIRS technology can be an auxiliary tool in the diagnosis of BD.

This study was performed with patients with suspected BD in emergency departments and intensive care units and was intended to evaluate the effectiveness of cerebral oximetry as an auxiliary diagnostic tool in patients with suspected BD.

ELIGIBILITY:
Inclusion Criteria:

1. All patients monitored and treated in the emergency department of intensive care units with a GCS score of 3 and evaluated as brain-dead at consultation with the Organ Transplantation Brain Death Committee on suspicion of BD
2. Aged over 18 years

Exclusion Criteria:

1. Cause of coma being undetermined
2. Lack of confirmation of brain injury being diffuse and irreversible
3. Central body temperature being lower than 32°C
4. Presence of a picture of hypotensive shock
5. Coma after drug effects and intoxications
6. Presence of metabolic, electrolyte or acid-alkaline disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential BD patients.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Basal ScO2 (Cerebral oxygen saturation) (%) | Measured at the beginning of 6 hours cerebral oximetry monitoring
End ScO2 (Cerebral oxygen saturation) (%) | Measured at the end of 6 hours cerebral oximetry monitoring
Mean ScO2 (Cerebral oxygen saturation) (%) | Measured during 6 hours cerebral oximetry monitoring
Min ScO2 (Cerebral oxygen saturation) (%) | Measured during 6 hours cerebral oximetry monitoring
Max ScO2 (Cerebral oxygen saturation) (%) | Measured during 6 h cerebral oximetry monitoring

SECONDARY OUTCOMES:
Decrease in ScO2 | Measured during 6 hours cerebral oximetry monitoring
  Difference between basal ScO2 and end ScO2

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes